CLINICAL TRIAL: NCT05502497
Title: Investigation of the Effect of Instrument Assisted Soft Tissue Mobilization Technique on Strength, Flexibility, Balance and Fascia and Fat Tissue Thickness in Healthy Individuals.
Brief Title: Investigation of the Effect of Instrument Assisted Soft Tissue Mobilization Technique on Fascia and Fat Tissue Thickness in Healthy Individuals.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Muhammed Usame TAS, Principal Investigator, Inonu University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ÜSAME TAŞ-002
Record Dates: First submitted 2022-08-13; First posted 2022-08-16 (Actual); Last update posted 2022-08-16 (Actual); Status verified 2022-08

CONDITIONS: Instrument-assisted Soft Tissue Mobilization; Flexibility; Fascia; Rehabilitation; Strength; Balance
MeSH Terms: interventions — Watchful Waiting

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Other): Which leg of the individuals will be treated will be determined by tossing a coin. After the toss, the right leg will be applied when the tail comes, and the left leg will be applied when it comes to the heads. The leg to be treated, the treatment group of the individuals; the other leg (the untreated leg) will form the control group of the individuals.
  Interventions: Other: Observational
- IASTM Treatment Group (Experimental): Which leg of the individuals will be treated will be determined by tossing a coin. After the toss, the right leg will be applied when the tail comes, and the left leg will be applied when it comes to the heads. The leg to be treated, the treatment group of the individuals; the other leg (the untreated leg) will form the control group of the individuals.
  Interventions: Other: IASTM Technique Application

INTERVENTIONS:
Other: Observational — No application will be made to the control group.
  Arms: Control Group
Other: IASTM Technique Application — Instrument-assisted soft tissue mobilization will be applied to the legs of the individuals to be treated with ultrasound gel for 2 minutes.
  Arms: IASTM Treatment Group

SUMMARY:
Instrument-assisted soft tissue mobilization (IASTM) technique can be used for non-pathological conditions as it has been shown in previous literature to affect flexibility and normal range of motion. The use of instrument-assisted soft tissue mobilization technique has been claimed to be an effective treatment in increasing tissue temperature, reducing adhesion to connective tissue and increasing collagen adaptation and increasing flexibility and normal range of motion. The instrument-assisted soft tissue mobilization technique works on the facial connective tissue in the body. This connective tissue contains "sheaths of collagen, which form the cavities and muscle divisions that mainly cover the organs." In some studies, they stated that instrument-assisted soft tissue mobilization increased perfusion, while in some studies they stated that instrument-assisted soft tissue mobilization increased blood circulation.

The frequency of ultrasonography (USG) examinations for the musculoskeletal system has increased over time with technological developments and USG has entered daily use in the evaluation of various pathological conditions belonging to this system thanks to its comparable results with MR examinations. The unique advantages of USG such as low cost, easy availability, relatively short examination time, and dynamic real-time comparison with the contralateral side have made it easier to use for musculoskeletal examinations.

The aim of this study is to investigate the effect of instrument-assisted soft tissue mobilization technique on strength, flexibility, balance, fascia and adipose tissue thickness in healthy individuals.

DETAILED DESCRIPTION:
In the study, iASTM will be applied to healthy individuals and the effect of this technique will be examined. Demographic information of individuals will be recorded; Individuals will be evaluated in detail in terms of muscle strength, flexibility, balance, and fascia and adipose tissue thickness.

The work plan; pre-treatment evaluation, followed by treatment, second evaluation immediately after the end of treatment and control evaluation (third evaluation) 1 hour after the end of treatment. The data collection period is planned as 1,5 year.

ELIGIBILITY:
Inclusion Criteria:

1. Consists of healthy individuals between the ages of 18-35,
2. No history of orthopedic injury (muscle, tendon, joint capsule, ligament damage or peripheral neuropathy) in the lower extremities in the last 1 year,
3. Being able to express himself without cognitive, cognitive and mental problems,
4. Voluntarily agree to participate in the study.

Exclusion Criteria:

1. Injury to any lower extremity between measurements during the treatment process,
2. Having a BMI over 25,
3. Surgery or arthritis in the last 1 year,
4. Not being able or unwilling to do the tests,
5. Not wanting to leave of their own accord.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-09-01 (Estimated); Study Completion 2022-10-01 (Estimated)

PRIMARY OUTCOMES:
Leg Muscle Strength Assessment | Pre-treatment assessment.
  The Vertical Jump Test will be used to evaluate the leg muscle strength of individuals.
Leg Muscle Strength Assessment | Second assessment immediately after the end of the 10-minute treatment.
  The Vertical Jump Test will be used to evaluate the leg muscle strength of individuals.
Leg Muscle Strength Assessment | Control evaluation 1 hour after the end of treatment (third evaluation).
  The Vertical Jump Test will be used to evaluate the leg muscle strength of individuals.
Flexibility Assessment | Pre-treatment assessment.
  The sit-and-reach Test will be used to assess the flexibility of individuals.
Flexibility Assessment | Second assessment immediately after the end of the 10-minute treatment.
  The sit-and-reach Test will be used to assess the flexibility of individuals.
Flexibility Assessment | Control evaluation 1 hour after the end of treatment (third evaluation).
  The sit-and-reach Test will be used to assess the flexibility of individuals.
Balance Assessment | Pre-treatment assessment.
  Stork Balance Test will be used to evaluate the balance of individuals.
Balance Assessment | Second assessment immediately after the end of the 10-minute treatment.
  Stork Balance Test will be used to evaluate the balance of individuals.
Balance Assessment | Control evaluation 1 hour after the end of treatment (third evaluation).
  Stork Balance Test will be used to evaluate the balance of individuals.
Fascia and Adipose Tissue Thickness Assessment | Pre-treatment assessment.
  Ultrasound device will be used to measure the thickness of individuals' fascia and adipose tissue.
Fascia and Adipose Tissue Thickness Assessment | Second assessment immediately after the end of the 10-minute treatment.
  Ultrasound device will be used to measure the thickness of individuals' fascia and adipose tissue.
Fascia and Adipose Tissue Thickness Assessment | Control evaluation 1 hour after the end of treatment (third evaluation).
  Ultrasound device will be used to measure the thickness of individuals' fascia and adipose tissue.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammed Üsame TAŞ, Lecturer, Principal Investigator — Inonu University
Locations (1):
- Inonu University, Malatya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No